CLINICAL TRIAL: NCT06771583
Title: Identification and Validation of Epigenetic Biomarkers of PMDD
Acronym: BIO
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00484410; 1R01MH135896 (NIH)
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: PMDD; Premenstrual Dysphoric Disorder (PMDD); Premenstrual Syndrome-PMS; Premenstrual Syndrome; Menstrual Cycle
Keywords: menstrual cycle; pms; luteal phase; womens health; reproductive health; reproductive mental health; epigenetics; dna methylation; premenstrual; pmdd; women
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Premenstrual Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Eligible participants that pass inclusion and exclusion criteria who do not have premenstrual mood symptoms.
- Premenstrual Dysphoric Disorder (PMDD): Eligible participants that pass inclusion and exclusion criteria who do have premenstrual mood symptoms. Symptoms must be severe enough to meet PMDD criteria.

SUMMARY:
This research is being done to examine epigenetic markers and mood changes across the menstrual cycle, particularly in premenstrual dysphoric disorder (PMDD). The investigators previously identified epigenetic biomarkers of postpartum depression, another reproductive affective disorder, and in this study aim to determine if these biomarkers also distinguish PMDD cases from healthy controls at different points in the menstrual cycle. By collecting biological samples (such as blood) and monitoring mood changes across the menstrual cycle, the investigators will be able to determine whether these epigenetic markers are associated with PMDD. The investigators plan to study these epigenetic markers during the follicular phase (roughly the first half of the menstrual cycle, from menses until ovulation) and the luteal phase (roughly the second half of the menstrual cycle, from ovulation to menses). The investigators will study this in two groups: 1) individuals who do NOT have premenstrual mood symptoms, and 2) individuals with premenstrual syndrome/premenstrual dysphoric disorder (PMS/PMDD). The results will provide a comprehensive view of the changes in these systems across the menstrual cycle. This will add to the investigators understanding of the mechanisms that may cause PMS/PMDD.

DETAILED DESCRIPTION:
Premenstrual dysphoric disorder (PMDD) is a reproductive affective disorder with impairing mood symptoms that emerge monthly in the premenstrual (luteal) phase of the menstrual cycle. Reproductive affective disorders, including PMDD and postpartum depression, can be conceptualized as disorders of hormone sensitivity - an abnormal brain response to ovarian hormone fluctuations. Epigenetic variations in prior studies by the investigators were prospectively predictive of postpartum depression risk with over 80% accuracy. Recently, in a cross-sectional cohort of 50 women with and without PMDD, this postpartum depression epigenetic biomarker distinguished PMDD cases from controls in the luteal phase, suggesting this may indicate sensitivity to reproductive hormone change. The primary aim of this study is to explore whether this epigenetic biomarker is a broad marker for hormone sensitivity, by assessing women (controls, PMDD) in both the follicular and luteal phases of the participant's menstrual cycles, using a repeated measures approach. A secondary aim is to examine whether the epigenetic biomarkers differ between women with PMDD who have responded to selective serotonin reuptake inhibitor (SSRI) treatment versus those who have failed SSRIs. SSRIs are the first-line treatment for PMDD, yet many PMDD patients do not respond to SSRIs. This study will assess DNA methylation in a cohort of women with PMDD and controls. The investigators will compare the epigenetic biomarker between controls and PMDD in the follicular and luteal phases. Within the PMDD group, the investigators will compare the biomarker between those who have responded to SSRI treatment and those who have not. Blood will be collected at home by participants using a dried blood spot collection system.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* regular menstrual cycles (24-35 days)
* age 18-50 years
* ability to give written informed consent

Exclusion Criteria:

* psychiatric medication use in the past 2 months;
* substance use disorder in the past 2 months (per MINI);
* lifetime history of psychotic disorder including schizophrenia, schizoaffective disorder, major depression with psychotic features (per MINI);
* history of psychiatric disorder other than PMDD in past year (per MINI);
* active suicidal ideation with plan or attempt in past 6 months (per MINI);
* steroid hormone or hormonal contraceptive use (except levonorgestrel as emergency contraceptive) in past 2 months;
* pregnancy in past 6 months;
* history of brain injury;
* current or history of endocrine disorder including uncontrolled diabetes or thyroid disease;
* BMI>40.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from Virginia, Washington DC, and Maryland (Baltimore area).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2030-02-15 (Estimated); Study Completion 2031-02-15 (Estimated)

PRIMARY OUTCOMES:
Presence of DNA Methylation Biomarkers (Comparing individuals with PMDD and controls) | From enrollment until study completion (approximately 3 months)
  In the luteal phase, DNA methylation variations at HP1BP3, TTC9B will distinguish controls from individuals with PMDD. In the follicular phase, DNA methylation variations at HP1BP3 and TTC9B will not distinguish controls from PMDD. The investigators will be collecting dried blood spots and assaying these epigenetic markers using various DNA methylation techniques.

SECONDARY OUTCOMES:
Presence of DNA Methylation Biomarkers (comparing history of SSRI treatment vs SSRI non response) | From enrollment until study completion (approximately 3 months)
  In the luteal phase, DNA methylation variations at HP1BP3, TTC9B will distinguish those with a history of SSRI treatment response versus SSRI non-response among women with PMDD. In the follicular phase, DNA methylation variations at HP1BP3, TTC9B will not distinguish those with a history of SSRI treatment response versus SSRI non-response among women with PMDD. Samples from which these assays are performed are from dried blood spots.
Epigenetic biomarkers associated with PMDD | From enrollment until study completion (approximately 3 months)
  Novel epigenetic biomarkers associated with PMDD will be identified using dried blood spots and associated methods and techniques for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Hantsoo, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Reproductive Mental Health Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The study information and a link to the screening form will be on this page following IRB approval. — https://tinyurl.com/rmhcstudies